CLINICAL TRIAL: NCT03639233
Title: Youth Epilepsy and Successful Self-Management Intervention
Acronym: YESS!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003214
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other): Intervention access
  Interventions: Behavioral: YESS!

INTERVENTIONS:
Behavioral: YESS! — Web based self-management education

SUMMARY:
This study is designed as a pilot test of the YESS! web-based intervention for adolescents with epilepsy. One hundred twenty participants will be given access to the intervention for a period of eight weeks. The investigators are testing the feasibility and acceptability of the the study procedures, measures and of the intervention itself. The study also evaluats the potential for impact on the users.

DETAILED DESCRIPTION:
YESS! is a web-based self management program developed to enhance the motivation and skills of youth with epilepsy.

This clinical trial uses a pre-test, post-test design where all consenting participants are given access to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age as above
* Epilepsy diagnosed by a physician
* Currently taking anti-seizure medications or use device
* Ability to understand and respond to questions about health and epilepsy
* Ability to utilize an internet based intervention website

Exclusion Criteria:

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting and enrollment procedures and | 8 weeks after getting access to the web intervention
  Measure the extent to which the recruitment and enrollment procedures meet the study aims in terms of number of participants log in to the intervention
Acceptability of intervention website users | 8 weeks after getting access to the web intervention
  and the extent to which users (study subjects) find the intervention easy to use, enjoyable to use, useful, engaging. Acceptability is a multifaceted and complex concept. As such it it is best examined as a system of interacting attributes.

SECONDARY OUTCOMES:
Participant Well-being | 8 weeks after getting access to the web intervention and 8 weeks after that.
  measures of overall well-being (EPOCH wellbeing meausre)
Participant Quality of Life | 8 weeks after getting access to the web intervention and 8 weeks after that.
  measure quality of life in epilepsy (QoLiE-10)
self-management behavior profile | 8 weeks after getting access to the web intervention and 8 weeks after that.
  measure the frequency of self management behaviors (taking medications, making clinic appointments, speaking with doctor/nurse/teacher) using a measure developed for this study
self-management motivation profile | 8 weeks after getting access to the web intervention and 8 weeks after that.
  measure the motivations (autonomous and extrinsic reasons for engaging in self management) using an adapted version of a standardized measure of motivation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Scal, MD MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
YESS! is a member of the Managing Epilepsy Well (MEW) and the associated shared database of deidentified participant records